CLINICAL TRIAL: NCT02688491
Title: A Multi-site, Open, Perspective Study of Prognostic Value and Benefit From Adjuvant Targeted Therapy of Stage III Clear Cell Renal Cell Carcinoma Based on a CpG-methylation-based Assay
Brief Title: A CpG-methylation-based Assay for Stratifying Stage III Clear Cell Renal Cell Carcinoma of Receiving Adjuvant Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Xi'an Jiaotong University (Other); Yantai Yuhuangding Hospital (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun-Hang Luo, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: [2016]015
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Renal Neoplasms; Targeted Molecular Therapy
MeSH Terms: conditions — Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Intervention group,sunitinib) (Experimental): Beginning 4-12 weeks following radical nephrectomy, patients receive sunitinib malate PO QD for 4 weeks
  Interventions: Drug: sunitinib
- B(observation group) (No Intervention): Patients with radical nephrectomy are observed without intervention

INTERVENTIONS:
Drug: sunitinib — The investigators randomly assign assay-defined high risk patients of stageIII ccRCC into intervention group and observation group. The intervention group should receive adjuvant targeted therapy while the control group deserve observation.
  Arms: A (Intervention group,sunitinib)

SUMMARY:
Whether patients with stage III clear cell renal cell carcinoma(ccRCC) should receive adjuvant targeted therapy or not is still on debate. The investigators invented a assay consisting of 5 CpGs: cg00396667（PITX1）, cg18815943 （FOXE3）, cg03890877（TWF2）, cg07611000 （EHBP1L1）and cg14391855（RIN1）that was successfully categorise patients with stage III clear cell renal cell carcinoma into high-risk and low-risk groups with Harzard Ratio(HR) of 4.93. Here the investigators randomly assign assay-defined high risk patients of locally advanced ccRCC into adjuvant targeted therapy group and observation group.Disease free survival and overall survival are the end points of observation.

DETAILED DESCRIPTION:
The investigators' CpG-methylation-based assay contains 5 CpGs: cg00396667（PITX1）, cg18815943 （FOXE3）, cg03890877（TWF2）, cg07611000 （EHBP1L1）and cg14391855（RIN1）. The investigators evaluate the CpG methylation status of surgical specimens using pyrosequencing and calculate their risk score[risk score=(0.0066×PITX1)+(0.0034×FOXE3)-(0.027×TWF2) -(0.018×EHBP1L1)-(0.03×RIN1)], risk score ≥-0.1 as assay-defined high risk status and risk score<-0.1 as assay-defined low risk status. The investigators randomly assign assay-defined high risk patients of stage III ccRCC into intervention group and control group. The intervention group should receive adjuvant targeted therapy while the control group deserve observation. Primary endpoint is the disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent has been obtained from the patient.
* With confirmed diagnosis of stage III clear cell renal cell carcinoma
* With moderate/good ECOG health rating (PS): 0-1 score.
* The patient receive no anti-cancer treatment before primary surgery.
* The patient receive radical operation for renal cancer with negative margin.

Exclusion Criteria:

* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.
* Pregnant woman or lactating woman.
* With contraindication to receive adjuvant targeted therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From the date of registration to up to10 years

SECONDARY OUTCOMES:
Overall survival | From the date of registration to up to10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hang Luo, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Undecided